- 16. Appendices
- 16.1. Study Information
- 16.1.9. Documentation of Statistical Methods

Statistical Analysis Plan, version 2.0, 09 October 2019



## STATISTICAL ANALYSIS PLAN

# STUDY TITLE:

A Phase I, Double-blind, Randomized, Placebo-controlled, Single Dose-escalation Study to Evaluate the Tolerability and Safety of Cytisine in Adult Smokers

Protocol Code: ACH-CYT-08

Type: Interventional, Phase I

EudraCT No.: 2018-003344-22

SAP Version: 2.0

Date: 09OCT2019

Supersedes version:

Date: 20MAY2019

Protocol Version 5.0

Sponsor: Achieve Life Sciences, Inc.

520 Pike Street, Suite 2250

Seattle, Washington, USA 98101

Phone: 604 736 3678 Fax: 604 736 3687

Clinical Pharmacology Unit:



## CONFIDENTIALITY DISCLAIMER

This document is confidential and is available for review to investigators, regulatory bodies and study audit personnel. No part of this document may be used, published, copied or otherwise disclosed without prior written authorization from Achieve Life Sciences, Inc.

Protocol: ACH-CYT-08 Version: 2.0 Date: 090CT2019




## 1. SIGNATURE PAGES

# 1.1. Clinical Pharmacology Unit's Representatives



# 1.2. Sponsor's Representatives





# 1.2. Sponsor's Representatives





## SUMMARY OF CHANGES OF THIS VERSION 2.0) VERSUS PREVIOUS VERSION (1.0)

Version 1.0 of this SAP was not implemented, as the study protocol was amended prior to database lock and final statistical analysis to include 3 additional dose cohorts. Version 2.0 of this SAP has incorporated analysis for dose cohorts 7 (24 mg), 8 (27 mg) and 9 (30 mg). No modifications to analysis plans have been made other than removing analysis of cotinine and 3-OH cotinine, as testing will not be conducted, per the Sponsor.

## 2. CONTENTS AND ABBREVIATIONS

## 2.1. Table of Contents

| 1. | SIGNA | SIGNATURE PAGES | | 2 |
|---|---|---|---|---|
| | 1.1.<br>1.2. | | PHARMACOLOGY UNIT'S REPRESENTATIVES | |
| 2. | CONTI | ENTS ANI | D ABBREVIATIONS | 4 |
| | 2.1.<br>2.2. | | CONTENTSBBREVIATIONS | |
| 3. | INTRO | DUCTIO | N | 8 |
| | 3.1.<br>3.2. | | OF CHANGES FROM PROTOCOL OR ITS AMENDMENTSG AND DELIVERABLES | |
| 4. | STUDY | OBJECT | TIVES | 8 |
| | 4.1.<br>4.2. | | Y | |
| 5. | STUDY | DESIGN | OVERVIEW | 9 |
| | 5.1.<br>5.2.<br>5.3.<br>5.4. | Number o | SIGN | 9<br>10 |
| 6. | STUDY | VARIAB | BLES | 10 |
| | 6.1.<br>6.2.<br>6.3. | PHARMACO | ORIABLES<br>ODYNAMIC VARIABLES<br>OKINETIC VARIABLES | 12 |
| 7. | DATA | REVIEW | / TRANSFORMATION | 12 |
| | 7.1.<br>7.2.<br>7.3. | ACCEPTAN | NAGEMENT<br>ICE OF DATA<br>NSFORMATION (CDISC) | 12 |
| 8. | STATI | STICAL N | METHODS | 13 |
| | 8.1. | ANALYSIS 8.1.1.<br>8.1.2.<br>8.1.3. | SETS Screening Analysis Set Safety Analysis Set Pharmacokinetic Analysis Set | 14<br>14 |



| | 8.2. | SUBJECT | DISPOSITION | 14 |
|---|---|---|---|---|
| | 8.3. | DEMOGE | RAPHIC AND OTHER BASELINE CHARACTERISTICS | 14 |
| | 8.4. | MEDICA | L AND SMOKING HISTORY | 14 |
| | 8.5. | Dosing. | | 15 |
| | 8.6. | Ркотос | OL DEVIATIONS | 15 |
| | 8.7. | SAFETY | Assessments | 15 |
| | | 8.7.1. | Adverse Events | |
| | | 8.7.2. | Laboratory Data | 16 |
| | | 8.7.3. | Vital Signs | 16 |
| | | 8.7.4. | | |
| | | 8.7.5. | | |
| | | 8.7.6. | Previous and Concomitant Medications | 17 |
| | 8.8. | PLASMA | CONCENTRATIONS | 17 |
| | 8.9. | | ACOKINETIC PARAMETERS | |
| | 8.10. | Dose-pf | ROPORTIONALITY | 18 |
| 9. | PRESE | ENTATIO | ON OF RESULTS | 18 |
| | 9.1. | STATIST | TICAL OUTPUT SPECIFICATION | 18 |
| | | 9.1.1. | | |
| | | 9.1.2.<br>9.1.3. | | |
| 10 | . REFE | RENCES | S | 23 |
| 11 | . APPEN | DICES. | | 24 |





#### 2.2. List of Abbreviations

ADAE Analysis Data Adverse Events

ADaM Analysis Data Model

ADEG Analysis Data Electrocardiogram

ADaMIG Analysis Data Model Implementation Guide

ADLB Analysis Data Laboratory

ADPC Analysis Data Pharmacokinetic Concentrations
ADPP Analysis Data Pharmacokinetic Parameters

ADSL Analysis Dataset, Subject-Level ADVS Analysis Data Vital Signs

AE Adverse Event

ALP Alkaline Phosphatase
ALT Alanine Aminotransferase

A<sub>mean</sub> Arithmetic mean

aPTT Activated Partial Thromboplastin Time

AST Aspartate Aminotransferase
ATC Anatomic Therapeutic Class
BLQ Below the Limit of Quantification

BMI Body Mass Index

C<sub>max</sub> Maximum Observed Plasma Concentration

CO Carbon Monoxide **CPK** Creatine Phosphokinase CR Clinically Relevant Creatinine Clearance  $Cr_{CL}$ Clinical Study Report **CSR** Coefficient of Variation CV% Diastolic Blood Pressure DBP **DSM** Data Safety Monitor **ECG** Electrocardiogram

GGT Gamma-Glutamyltransferase GLP Good Laboratory Practice

G<sub>mean</sub> Geometric mean

hCG Human Chorionic Gonadotropin HIV Human Immunodeficiency Virus INR International Normalized Ratio

LC-MS/MS Liquid Chromatography with Tandem Mass Spectrometry

LDH Lactate Dehydrogenase
LLOQ Lower Limit of Quantification
MCH Mean Corpuscular Hemoglobin

MCHC Mean Corpuscular Hemoglobin Concentration

MCV Mean Corpuscular Volume

MedDRA Medical Dictionary for Regulatory Activities

NCR Not Clinically Relevant
NMR Nicotine Metabolite Ratio
PI Principal Investigator
PT MedDRA Preferred Term

RBC Red Blood Cell

Protocol: ACH-CYT-08 Version: 2.0

Date: 09OCT2019



| RDW-CV | Coefficient Variation of the Red Cell Distribution Width |
|-----------|-------------------------------------------------------------|
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SBP | Systolic Blood Pressure |
| SD | Standard Deviation |
| SOC | MedDRA System Organ Class |
| TEAE | Treatment-Emergent Adverse Events |
| TFLs | Tables, figures and listings |
| $T_{max}$ | Time of Occurrence of Maximum Observed Plasma Concentration |
| ULOQ | Upper Limit of Quantification |
| WBC | White Blood Cell |



#### 3. INTRODUCTION

This Statistical Analysis Plan (SAP) presents the details of the analysis and presentation of the safety and pharmacokinetic (PK) results for Clinical Study ACH-CYT-08.

The analyses described are based on the Clinical Study Protocol (CSP) version 5.0, dated 07MAY2019 [1].

This SAP will be finalized and approved by the Achieve Life Sciences (Achieve) and s representatives prior to the planned database lock and unblinding of study treatment assignment code. Any deviations from this SAP will be described in detail and justified in the Clinical Study Report (CSR). If additional analyses are required to complement the analyses planned in the SAP, they may be performed and will be identified in the Clinical Study Report (CSR).

# 3.1. Summary of Changes from Protocol or Its Amendments

There are no changes from the protocol or its amendments.

## 3.2. Reporting and Deliverables

The CSR will be written using the Achieve's template. Tables, Figures and Listings (TFLs) will be prepared as described in the TFL shells within this SAP. In-text Tables and Figures will be included in the main body of the CSR. After review by the Sponsor, the TFLs will be finalized.

Before performing the analysis, all data collected will be integrated into a common repository, using SAS 9.4 (SAS Institute Inc, Cary, NC, USA). Derived analysis datasets will be generated in accordance to CDISC. ADaM compliant datasets will be delivered to the Sponsor.

## 4. STUDY OBJECTIVES

## 4.1. Primary

To assess the tolerability and safety of cytisine as a single oral dose.

# 4.2. Secondary

To define the  $C_{max}$  levels associated to the occurrence of dose-limiting adverse events.



#### 5. STUDY DESIGN OVERVIEW

## 5.1. Study Design

This was a single-center, double-blind, randomized, placebo-controlled, single dose-escalation, Phase 1 clinical study conducted in male or female adults who were in good general health and were current daily cigarette smokers, under fasting conditions.

Nine dose levels were pre-planned under version 5.0 of Protocol ACH-CYT-08: 6 mg, 9 mg, 12 mg, 15 mg, 18 mg, 21 mg, 24 mg, 27 mg and 30 mg. The starting dose was 6 mg cytisine (single oral dose) in Cohort 1. The study was escalated up to the cytisine dose of 30 mg in Cohort 9 without showing any of the predefined stopping criteria. Within each dose level, subjects were randomly assigned to receive a single oral dose of cytisine or placebo in a 3:1 ratio (6 cytisine:2 placebo).

Upon completion of a cohort, a safety review was performed by the Principal Investigator (PI) and two independent Data Safety Monitors (DSMs) on unblinded data. The PI and DSMs conjointly decided whether dose escalation into the next cohort was to be allowed.

Table 1 presents an overview of study design.

Treatment Period in Each Cohort Screening Admission Confinement Follow-up Escalation to Next Cohort Decision D -28 to D -1 D 0 D 1 D2 D 5/D6 Eligibility Eligibility Check Single-dose Discharge Safety Review Evaluation Administration Randomization 6 cytisine : 2 placebo

Figure 1. Study Diagram:

#### 5.2. Number of Subjects

**Adverse Events Monitoring** 

The study protocol defined a sample size of 8 subjects per cohort, which is consistent with standard practice in early-phase clinical trials with similar study objectives.

Considering that 9 cohorts were pre-planned, a total of 72 subjects was estimated for enrollment.

Protocol: ACH-CYT-08 Version: 2.0 Date: 09OCT2019



#### **5.3.** Number of Clinical Sites

This was a single center clinical trial.

# 5.4. Method of Assigning Subjects to Treatments

Using SAS® 9.4, a computer-generated block-wise randomization list adequate for placebo-controlled studies was prepared by the Programming & Biostatistics Department of At each cohort, 6 subjects were randomly assigned to receive cytisine and 2 subjects randomized to receive placebo.

Upon confirmation that all eligibility criteria are met on Day 0, subjects were sequentially assigned a randomization number. The randomization number was provided to the unblinded Pharmacist on site and defined the treatment to which subjects were allocated (test or placebo) per the randomization list.

#### 6. STUDY VARIABLES

## 6.1. Safety variables

- Drug exposure
- Adverse events:
  - Reported Term
  - MedDRA SOC coding
  - MedDRA PT coding
  - Start date
  - Start time
  - End date
  - End time
  - Seriousness
  - Severity:
    - Mild
    - Moderate
    - Severe
  - Relationship (causality):
    - not related
    - unlikely
    - possible
    - probable
    - definite
  - Action taken
    Outcome
- Clinical laboratory evaluations:
  - Biochemistry:
    - aspartate aminotransferase (AST)
    - alanine aminotransferase (ALT)


Protocol: ACH-CYT-08 Version: 2.0 Date: 09OCT2019



- gamma-glutamyltransferase (GGT)
- lactate dehydrogenase (LDH)
- alkaline phosphatase (ALP)
- creatine phosphokinase (CPK)
- creatinine
- estimated creatinine clearance (CR<sub>CL</sub>)
- urea
- sodium
- potassium
- calcium
- glucose
- total cholesterol
- triglycerides
- albumin
- total protein
- uric acid
- direct bilirubin
- indirect bilirubin
- total bilirubin
- Hematology:
  - hemoglobin
  - hematocrit
  - hypochromic red blood cell
  - red blood cell (RBC) count
  - mean corpuscular volume (MCV)
  - mean corpuscular hemoglobin (MCH)
  - mean corpuscular hemoglobin concentration (MCHC)
  - coefficient variation of the red cell distribution width (RDW-CV)
  - total white blood cell (WBC) count
  - neutrophils
  - eosinophils
  - lymphocytes
  - monocytes
  - basophils
  - platelet count
- Coagulation:
  - prothrombin rate
  - prothrombin time international normalized ratio (INR)
  - activated partial thromboplastin time (aPTT)
- Urinalysis:
  - pH
  - specific gravity
  - protein
  - hemoglobin
  - glucose
  - ketones
  - bilirubin
  - nitrites



- urobilinogen
- microscopy
- Drugs of abuse test:
  - cannabinoids
  - opiates
  - cocaine
  - amphetamines
  - benzodiazepines
- Serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test
- Urine beta-hCG pregnancy test
- Ethanol breath test
- Vital signs:
  - Systolic blood pressure (SBP)
  - Diastolic blood pressure (DBP)
  - Pulse rate
  - Body temperature
- Physical examination
- 12-lead Electrocardiogram (ECG)
- CO

## 6.2. Pharmacodynamic variables

None.

#### 6.3. Pharmacokinetic Variables

- Plasma concentrations of cytisine
- Maximum observed plasma concentration post dose, directly obtained from the observed cytisine concentration versus time profile (C<sub>max</sub>)
- Time of occurrence of  $C_{max}$  ( $T_{max}$ )

#### 7. DATA REVIEW / TRANSFORMATION

## 7.1. Data Management

Data handling will be conducted in accordance with the Clinical Data Management section of the CSP and the Data Management Plan developed by study.

## 7.2. Acceptance of Data

TFLs may start being programmed prior to, or during, the course of the trial. However, the programming of analysis datasets (ADS) and TFLs will only be finished and quality-controlled after database soft lock and unblinding of the data. Only audited cytisine plasma concentration data released by the Bioanalytical Laboratory will be used



for programming the final pharmacokinetic ADS and TFLs.

# 7.3. Data Transformation (CDISC)

Before performing the statistical analysis, all data collected (multiple sources) will be integrated into a common repository, using SAS® 9.4.

For standardization and regulatory submission purposes, all data will be transformed according to Clinical Data Interchange Standards Consortium (CDISC):

- Study Data Tabulation Model (SDTM) version 1.4 or later;
- Study Data Tabulation Model Implementation Guide (SDTMIG) version 3.2 or later;
- The following analysis datasets will be generated (Analysis Data Model [ADaM] version 2.1; Analysis Data Model Implementation Guide [ADaMIG], version 1.1) to support the results and ease the programming activities during the statistical analysis:
  - Subject-Level Analysis Dataset (ADSL)
  - Analysis Data Adverse Events (ADAE)
  - Analysis Data Electrocardiogram (ADEG)
  - Analysis Data Vital Signs (ADVS)
  - Analysis Data Laboratory (ADLB)
  - Analysis Data Pharmacokinetic Concentrations (ADPC)
  - Analysis Data Pharmacokinetic Parameters (ADPP)

#### 8. STATISTICAL METHODS

The statistical analysis and TFLs will be done using SAS® for version 9.4.

PK parameters for cytisine ( $C_{max}$  and  $T_{max}$ ) will be estimated using non-compartmental analysis (NCA) in Phoenix<sup>®</sup> WinNonlin<sup>®</sup> version 8.1 (Pharsight Corp., Mountain View, CA).

Summaries of demographics, baseline characteristics and safety endpoints will be provided for the Safety Analysis Set, defined as all subjects who received a single dose of cytisine or placebo.

Unless otherwise indicated, numerical variables will be summarized using: number of observations (n), arithmetic mean, standard deviation, coefficient of variation (CV%), median and range (minimum and maximum). Categorical variables will be summarized with number of subjects and percentage within a treatment (dose level). Descriptive statistics will be presented with the same precision as the original data, i.e, the same number of decimals or significant digits. T<sub>max</sub> is stated with the same number of significant digits as the actual sampling time. Baseline for post-dose assessments is defined as the last observation recorded before dose. Summaries will be provided for each dose level/treatment (Placebo; 6.0 mg cytisine; 9.0 mg cytisine, etc.). Unless otherwise indicated, no statistical comparisons between the cohorts are planned.

Unscheduled measurements will be listed in the individual data listings. With the 

exception of baseline or unscheduled measurements performed due to an error at the scheduled measurement (e.g. equipment failure), unscheduled measurements will be excluded from the descriptive statistical analysis.

No imputation of missing data will be done, except for missing dates and/or times required for the calculation of AEs' time to onset and duration (e.g. see Section 8.7.1) and for plasma concentrations below the lower limit of quantification (LLOQ) (see Section 8.8).

Assessments for trends in dose-limiting adverse events or  $C_{max}$  levels in relationship to BMI categories/levels and baseline Nicotine Metabolite Ratio (NMR) may be explored.

## 8.1. Analysis Sets

## 8.1.1. Screening Analysis Set

The Screening Analysis Set is defined as all subjects who give written informed consent and have entered screening. Analyses will be restricted to presentation of baseline data and reasons for non-participation as contrasted to those enrolled and received study drug.

## 8.1.2. Safety Analysis Set

The Safety Analysis Set is defined as all enrolled subjects who were administered the single dose of study drug.

## 8.1.3. Pharmacokinetic Analysis Set

The Pharmacokinetic Analysis Set is defined as all subjects who received a dose of cytisine and have evaluable pharmacokinetic data.

## 8.2. Subject Disposition

The number and percentage of subjects who meet study analysis set requirements will be presented, along with number and percentage of subjects who prematurely withdrew. Reasons for withdrawal will be included.

## 8.3. Demographic and Other Baseline Characteristics

Subjects demographic data (except date of birth) and other baseline characteristics will be collected at screening and will be listed and summarized descriptively for all subjects by treatment and overall. The data in the summary will include age (years), sex, race, height (cm), weight (kg) and body mass index (BMI, kg/m²).

## 8.4. Medical and Smoking History

Medical history will be collected at screening and coded using the MedDRA dictionary version 21.1 or higher. Coding includes system organ class (SOC) and preferred term


(PT). Medical history events will be listed for all subjects. Frequencies of medical history events will be presented by SOC and PT, by treatment and overall.

Smoking history will be collected at screening and will be listed and summarized descriptively for all subjects by treatment and overall. The data in the summary will include duration (years) of smoking, average number of cigarettes smoked per day during the last 30 days, whether subject ever attempted to quit smoking (Yes, No). In addition, the following will be summarized for subjects who had ever attempted to quit smoking: number of previous quit attempts, time (months) since most recent quit attempt and smoking cessation treatments used. The summary of smoking cessation treatments will report the number and percentage of subjects that used each treatment, as well as the number (%) of subjects that used any prior nicotine replacement therapy (i.e., used nicotine gum or nicotine patch or nicotine nasal spray or nicotine inhaler).

Expired CO level (ppm) will be measured at screening. These data will be listed for all subjects and summarized for all subjects by treatment and overall.

## 8.5. Dosing

Study product administration dates and times will be listed.

#### **8.6.** Protocol Deviations

Protocol deviations will be listed.

## 8.7. Safety Assessments

#### 8.7.1. Adverse Events

Clinically significant abnormalities will be reported as AEs. Adverse events will be coded using the MedDRA dictionary version 21.1 or higher. Coding includes system organ class (SOC) and preferred term (PT). The following information recorded or computed is used for the description of the AEs: reported Term; SOC and PT by MedDRA coding; start date, start time, end date and end time; seriousness; severity (intensity); relationship (causality); action taken; outcome. AE duration and time to AE onset will be derived and presented in the subject data listings.

TEAEs will be presented by dose level. TEAEs are defined as AEs not present prior to administration of investigational product, or AEs present before administration of investigational product that worsen after the subject received the investigational product. A separate listing of SAEs will be presented, if applicable. Frequencies of TEAEs will be presented by SOC and PT, by Test product and placebo and overall.

TEAEs of which the relationship to the test drug was classified as 'possible', 'probable' and 'definite' will be regarded as "related", while TEAEs that are classified as 'not related' or 'unlikely' will be regarded as "not related".

Frequencies of TEAEs will also be reported by severity class (Mild, Moderate, or

Severe) and by investigational product and dose, for all causalities and for "related" events.

#### 8.7.2. Laboratory Data

Individual laboratory test data will be listed. A listing of the values outside the prespecified ranges will be flagged ("H" - high or "L" - low) and classified regarding clinical relevance.

A decision regarding whether a result outside the reference range is of clinical significance or not was made by the clinical investigator and reported and annotated accordingly. Clinically significant abnormalities occurring during the study will be recorded as AEs.

The reference ranges for the site's laboratory parameters will also be entered in the database and filed in the Investigator site file.

#### 8.7.3. Vital Signs

Continuous vital signs monitoring (heart rate, respiratory rate and pulse oximetry) will be performed from pre-dose up to 6 hours post-dose. No listing of these data will be provided. Clinically relevant abnormalities during the period of continuous monitoring will be reported as AEs.

Vital signs (systolic blood pressure (SBP), diastolic blood pressure (DBP), pulse rate and body temperature) will be assessed at the following time points: Day 1 pre-dose, again at approximately 2, 4 and 6 hours post-dose on Day 1, and at discharge on Day 2.

Individual vital signs results will be listed. Out of range values will be flagged ("H" - high or "L" - low) and classified regarding clinical relevance. Clinically relevant abnormalities will be reported as AEs.

**Table 2. Vital Signs: Reference Values** 

| | Reference Values |
|------------------------|-----------------------------------|
| SBP (mmHg) | $90 \le SBP \le 120 \text{ mmHg}$ |
| DBP (mmHg) | $60 \le DBP \le 90 \text{ mmHg}$ |
| Heart Rate (beats/min) | 60 to 100 beats/min |
| Body Temperature (°C) | 35.5 to 37.5 °C |

## 8.7.4. Electrocardiograms

The ECG results will be listed per subject as "normal" or "abnormal". All abnormalities will be classified in terms of clinical relevance (CR, NCR). Clinically relevant abnormalities will be reported as AEs.

## 8.7.5. Physical Examinations

Clinically relevant changes from screening in physical examination will be reported as AEs.

## 8.7.6. Previous and Concomitant Medications

All other medications used will be listed as concomitant medications.

Previous/Concomitant medications will be coded according Anatomical Therapeutic Chemical (ATC) classification system.

#### 8.8. Plasma Concentrations

will carry out the determination of plasma levels of cytisine in accordance with the applicable principles of Good Laboratory Practices (GLP), using a previously validated LC-MS/MS analytical method. The pre-planned lower limit of quantification (LLOQ) is 1 ng/mL and the upper limit of quantification (ULOQ) is 400 ng/mL.

Individual (per subject) and mean plasma concentration versus time profiles will be presented for both linear and semi-logarithmic scales. Graphic presentation of individual data will be based on actual blood sampling time, except for pre-dose sampling time which will be assumed as t0.

Descriptive statistics (number of subjects, geometric mean, arithmetic mean, SD, CV%, median, minimum and maximum) of the plasma concentrations will be presented for each time point. Concentrations below the LLOQ will be taken as missing for the calculation of geometric mean and replaced by zero for calculation of the remaining summary statistics.

The pre-dose blood samples were to be collected within 30 minutes prior to dosing. The post-dose blood samples were to be collected within +/-2 minutes from the scheduled sampling time. The clock time was to be recorded and reported for all blood draws and all subjects. A deviation greater than +/-2 minutes will be reported as a protocol deviation and its cause will be recorded.

#### 8.9. Pharmacokinetic Parameters

Pharmacokinetic parameters will be estimated from the plasma concentration versus time profiles for all subjects in the pharmacokinetic analysis set.

Pharmacokinetic parameter  $C_{max}$  will be calculated as the maximum observed plasma concentration (ng/mL) and  $T_{max}$  will be the time to occurrence of maximum plasma concentration (h).

Individual PK parameters and descriptive statistics (number of subjects, arithmetic and geometric mean, SD, CV%, median, minimum value, and maximum value) will be presented by Cytisine Dose Level. For C<sub>max</sub> the 90% CI of the mean will also be 

estimated. If for more than  $\frac{1}{3}$  of the subjects no reliable PK parameter could be determined, only the minimum and maximum values will be presented for that parameter and all other descriptive statistics will be omitted. Missing PK parameter data will not be imputed.

## 8.10. Dose-proportionality

Linear-dose proportionality of  $C_{max}$  after oral administration of Cytisine 6 mg, 9 mg, 12 mg, 15 mg, 18 mg, 21 mg, 24 mg, 27 mg and 30 mg will be assessed by using an exponential regression model that measures the degree of nonlinear proportionality. The relationship is written as a power function:  $y = \alpha * dose^{\beta}$ , where y denotes the pharmacokinetic parameter being analyzed ( $C_{max}$ ),  $\alpha$  is a constant and  $\beta$  is the proportionality constant. Linearization of this relationship gives:

$$\log (y) = \log (\alpha) + \beta * \log (dose).$$

The relationship is dose proportional when  $\beta=1$  (linear pharmacokinetics) or considered to be dose dependent (non-linear pharmacokinetics) when  $\beta \neq 1$ . The exponent of the power function fitted to the individual  $C_{max}$  values and 95% CI will be assessed.

## 9. PRESENTATION OF RESULTS

#### 9.1. Statistical Output Specification

The summary tables will be generated as Rich Text Files (\*.rtf) from SAS<sup>®</sup> and compiled in a document, to be considered as Section 14 (Tables, Figures and Graphs Referred to But Not Included in the Text) of the CSR.

Tables and Figures for direct insertion in the body of the CSR, will also be generated as \*.rtf files. In-text tables and figures will preferably be prepared in portrait format. Listings will preferably be prepared in landscape format.

The planned TFLs for the CSR are listed below.

## 9.1.1. In-text Tables and Figures

## For CSR Synopsis:

Tables and/or Figures to be inserted in the synopsis of the CSR will be decided at the time of writing the CSR.

#### For CSR Body Text:

The planned tables and figures for CSR body text are listed below. Other relevant tables and/or figures may be presented in the final CSR body text. Thus, the placement and numbering presented is indicative and may deviate from the placement and numbering in the final CSR body text.



| <b>In-text Tables</b> | Title |
|---|---|
| Table A | Study Flow-Chart (to be captured from the CSP) |
| Table B | Identity of Investigational Products |
| Table C | Treatment Assignment |
| Table D | Subjects Disposition |
| Table E | Major Protocol Deviations |
| Table F.1 | Demographic Data – Safety Analysis Set |
| Table F.2 | Smoking History – Safety Analysis Set |
| Table F.3 | Baseline CO – Safety Analysis Set |
| Table G.1 | Treatment Emergent Adverse Events – All Causalities |
| Table G.2 | Treatment Emergent Adverse Events – Related |
| Table H | Cytisine: C <sub>max</sub> and T <sub>max</sub> Following Administration of Cytisine (6 |
| | mg, 9 mg, 12 mg, 15 mg, 18 mg, 21 mg, 24 mg, 27 mg and 30 |
| | mg) |
| Table I | Cytisine: Dose Proportionality of C <sub>max</sub> |

| <b>In-text Figures</b> | Legend |
|---|---|
| Figure A | Cytisine: Arithmetic Mean Plasma Concentration Versus Time |
| | Profile Following Administration of Cytisine (6 mg, 9 mg, 12 |
| | mg, 15 mg, 18 mg, 21 mg, 24 mg, 27 mg and 30 mg) – Linear |
| | Scale. |
| Figure B | Cytisine: Arithmetic Mean Plasma Concentration Versus Time |
| | Profile Following Administration of Cytisine (6 mg, 9 mg, 12 |
| | mg, 15 mg, 18 mg, 21 mg, 24 mg, 27 mg and 30 mg) – Semi- |
| | Logarithmic Scale |
| Figure C | Cytisine: Dose Proportionality of C <sub>max</sub> |
| Figure D | Cytisine: Boxplots of C <sub>max</sub> as a Function of Dose |

| End-of-Text | Title |
|---|---|
| Tables | |
| 14.1 DEMOGRA | 14.1 DEMOGRAPHIC DATA |
| 14.1.1 | Demographic Data – Safety Analysis Set |
| 14.1.2 | Smoking History – Safety Analysis Set (Part I) |
| 14.1.3 | Smoking History – Safety Analysis Set (Part II) |
| 14.1.4 | Smoking History – Expired CO at Screening |
| 14.1.5 | Medical History – Safety Analysis Set |
| 14.2 SAFETY D | 14.2 SAFETY DATA |
| 14.2.1 | Treatment Emergent Adverse Events |
| 14.2.1.1 | Adverse Events Leading to Discontinuation or Withdrawal |
| 14.2.1.2 | Listings of Serious Adverse Events |
| 14.2.1.3 | Summary of Treatment Emergent Adverse Events – All |
| | Causalities |
| 14.2.1.4 | Summary of Treatment Emergent Adverse Events - Related |
| 14.2.1.5 | Summary of Treatment Emergent Adverse Events by Severity – |




| | All Causalities |
|---|---|
| 14.2.1.6 | Summary of Treatment Emergent Adverse Events by Severity – |
| | Related |
| | ACOKINETIC DATA |
| 14.3.1 | Deviations from Blood Sampling Schedule |
| 14.3.1.1 | Deviations from Blood Sampling Schedule |
| 14.3.1.2 | Missing Blood Samples |
| 14.3.2 | Plasma Concentrations |
| 14.3.2.1 | Cytisine 6 mg: Individual Data and Descriptive Statistics of |
| | Plasma Concentrations |
| 14.3.2.2 | Cytisine 9 mg: Individual Data and Descriptive Statistics of |
| 11222 | Plasma Concentrations |
| 14.3.2.3 | Cytisine 12 mg: Individual Data and Descriptive Statistics of |
| 14224 | Plasma Concentrations |
| 14.3.2.4 | Cytisine 15 mg: Individual Data and Descriptive Statistics of |
| 14225 | Plasma Concentrations |
| 14.3.2.5 | Cytisine 18 mg: Individual Data and Descriptive Statistics of Plasma Concentrations |
| 14.3.2.6 | Cytisine 21 mg: Individual Data and Descriptive Statistics of |
| 14.3.2.0 | Plasma Concentrations |
| 14.3.2.7 | Cytisine 24 mg: Individual Data and Descriptive Statistics of |
| 14.3.2.7 | Plasma Concentrations |
| 14.3.2.8 | Cytisine 27 mg: Individual Data and Descriptive Statistics of |
| 11.3.2.0 | Plasma Concentrations |
| 14.3.2.9 | Cytisine 30 mg: Individual Data and Descriptive Statistics of |
| | Plasma Concentrations |
| 14.3.3 | Pharmacokinetic Parameters |
| 14.3.3.1 | Cytisine 6 mg: Individual Data and Descriptive Statistics of |
| | Pharmacokinetic Parameters |
| 14.3.3.2 | Cytisine 9 mg: Individual Data and Descriptive Statistics of |
| | Pharmacokinetic Parameters |
| 14.3.3.3 | Cytisine 12 mg: Individual Data and Descriptive Statistics of |
| | Pharmacokinetic Parameters |
| 14.3.3.4 | Cytisine 15 mg: Individual Data and Descriptive Statistics of |
| | Pharmacokinetic Parameters |
| 14.3.3.5 | Cytisine 18 mg: Individual Data and Descriptive Statistics of |
| 11226 | Pharmacokinetic Parameters |
| 14.3.3.6 | Cytisine 21 mg: Individual Data and Descriptive Statistics of |
| 14227 | Pharmacokinetic Parameters |
| 14.3.3.7 | Cytisine 24 mg: Individual Data and Descriptive Statistics of |
| 1/220 | Pharmacokinetic Parameters Cyticing 27 mg: Individual Date and Descriptive Statistics of |
| 14.3.3.8 | Cytisine 27 mg: Individual Data and Descriptive Statistics of |
| 14.3.3.9 | Pharmacokinetic Parameters Cyticine 30 mg: Individual Data and Descriptive Statistics of |
| 14.3.3.9 | Cytisine 30 mg: Individual Data and Descriptive Statistics of Pharmacokinetic Parameters |
| | r narmacokinetic rarameters |



| End-of-Text | Title |
|---|---|
| Figures 14.3 PHARMACOKINETIC DATA | |
| 14.3.4 | Cytisine Plasma Concentration-Time Profiles of All Subjects |
| 14.3.4.1 | Cytisine 6 mg: Plasma Concentration-Time Profiles of All |
| 14.3.4.1 | Subjects |
| 14.3.4.2 | Cytisine 9 mg: Plasma Concentration-Time Profiles of All |
| 17.5.7.2 | Subjects |
| 14.3.4.3 | Cytisine 12 mg: Plasma Concentration-Time Profiles of All |
| 11.5.1.5 | Subjects |
| 14.3.4.4 | Cytisine 15 mg: Plasma Concentration-Time Profiles of All |
| | Subjects |
| 14.3.4.5 | Cytisine 18 mg: Plasma Concentration-Time Profiles of All |
| | Subjects |
| 14.3.4.6 | Cytisine 21 mg: Plasma Concentration-Time Profiles of All |
| | Subjects |
| 14.3.4.7 | Cytisine 24 mg: Plasma Concentration-Time Profiles of All |
| | Subjects |
| 14.3.4.8 | Cytisine 27 mg: Plasma Concentration-Time Profiles of All |
| 11212 | Subjects |
| 14.3.4.9 | Cytisine 30 mg: Plasma Concentration-Time Profiles of All |
| | Subjects |
| 1425 | |
| 1 1 / 4 / | L'vitiging A withmotic Moon Plagma Concentration Time |
| 14.3.5 | Cytisine Arithmetic Mean Plasma Concentration-Time<br>Profiles |
| 14.3.5.1 | Profiles |
| | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus |
| 14.3.5.1 | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale |
| 14.3.5.1 | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus |
| 14.3.5.1<br>14.3.5.2<br>14.3.5.3 | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale |
| 14.3.5.1 | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus |
| 14.3.5.1<br>14.3.5.2<br>14.3.5.3<br>14.3.5.4 | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale |
| 14.3.5.1<br>14.3.5.2<br>14.3.5.3 | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus |
| 14.3.5.1<br>14.3.5.2<br>14.3.5.3<br>14.3.5.4<br>14.3.5.5 | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale |
| 14.3.5.1<br>14.3.5.2<br>14.3.5.3<br>14.3.5.4 | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus |
| 14.3.5.1<br>14.3.5.2<br>14.3.5.3<br>14.3.5.4<br>14.3.5.5<br>14.3.5.6 | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale |
| 14.3.5.1<br>14.3.5.2<br>14.3.5.3<br>14.3.5.4<br>14.3.5.5 | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus |
| 14.3.5.1<br>14.3.5.2<br>14.3.5.3<br>14.3.5.4<br>14.3.5.5<br>14.3.5.6<br>14.3.5.7 | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale |
| 14.3.5.1<br>14.3.5.2<br>14.3.5.3<br>14.3.5.4<br>14.3.5.5<br>14.3.5.6 | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale |
| 14.3.5.1<br>14.3.5.2<br>14.3.5.3<br>14.3.5.4<br>14.3.5.5<br>14.3.5.6<br>14.3.5.7 | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale |
| 14.3.5.1<br>14.3.5.2<br>14.3.5.3<br>14.3.5.4<br>14.3.5.5<br>14.3.5.6<br>14.3.5.7<br>14.3.5.8 | Profiles Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale |
| 14.3.5.1<br>14.3.5.2<br>14.3.5.3<br>14.3.5.4<br>14.3.5.5<br>14.3.5.6<br>14.3.5.7<br>14.3.5.8 | Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 18 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 18 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 18 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 18 mg: Arithmetic Mean Plasma Concentration Versus |
| 14.3.5.1<br>14.3.5.2<br>14.3.5.3<br>14.3.5.4<br>14.3.5.5<br>14.3.5.6<br>14.3.5.7<br>14.3.5.8<br>14.3.5.9 | Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 6 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 9 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 12 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Linear Scale Cytisine 15 mg: Arithmetic Mean Plasma Concentration Versus Time Profile – Semi-Logarithmic Scale Cytisine 18 mg: Arithmetic Mean Plasma Concentration Versus |



| | Time Profile – Linear Scale |
|-----------|-------------------------------------------------------------|
| 14.3.5.12 | Cytisine 21 mg: Arithmetic Mean Plasma Concentration Versus |
| | Time Profile – Semi-Logarithmic Scale |
| 14.3.5.13 | Cytisine 24 mg: Arithmetic Mean Plasma Concentration Versus |
| | Time Profile – Linear Scale |
| 14.3.5.14 | Cytisine 24 mg: Arithmetic Mean Plasma Concentration Versus |
| | Time Profile – Semi-Logarithmic Scale |
| 14.3.5.15 | Cytisine 27 mg: Arithmetic Mean Plasma Concentration Versus |
| | Time Profile – Linear Scale |
| 14.3.5.16 | Cytisine 27 mg: Arithmetic Mean Plasma Concentration Versus |
| | Time Profile – Semi-Logarithmic Scale |
| 14.3.5.17 | Cytisine 30 mg: Arithmetic Mean Plasma Concentration Versus |
| | Time Profile – Linear Scale |
| 14.3.5.18 | Cytisine 30 mg: Arithmetic Mean Plasma Concentration Versus |
| | Time Profile – Semi-Logarithmic Scale |

# 9.1.2. List of Subject Data Listings (Section 16.2 of CSR)

# 9.1.3.

The following data listings will be produced, to form Section 16.2. Subject Data Listings of the CSR:

| Listing No. | Title |
|---|---|
| 16.2 SUBJECT DATA LISTINGS | |
| 16.2.1 | Subject Disposition |
| 16.2.1.1 | Subject Disposition: Eligibility and Randomization |
| 16.2.2 | Protocol Deviations |
| 16.2.2.1 | Blood Sampling Time Deviations |
| 16.2.2.2 | Other Protocol Deviations |
| 16.2.3 | Demographic Data and Other Baseline Data |
| 16.2.3.1 | Demographic Data |
| 16.2.3.2 | Fertility/Contraception |
| 16.2.3.2.1 | Female Fertility/Contraception |
| 16.2.3.2.2 | Male Fertility/Contraception |
| 16.2.3.3 | Medical History at Screening |
| 16.2.3.4 | Smoking History at Screening |
| 16.2.3.5 | Expired CO at Screening |
| 16.2.3.6 | Drugs of Abuse and Ethanol |
| 16.2.3.7 | Previous Medication |
| 16.2.4 | Compliance |
| 16.2.4.1 | Investigational Product Administration |
| 16.2.5 | Adverse Event Listings (Each Subject) |
| 16.2.5.1 | Serious Adverse events (Part I) |
| 16.2.5.2 | Serious Adverse events (Part II) |
| 16.2.5.3 | Serious Adverse events (Part III) |
| 16.2.5.4 | Serious Adverse events (Part IV) |
| 16.2.5.5 | Serious Adverse events (Part V) |
| 16.2.5.6 | Treatment-Emergent Adverse Events |




| 16.2.5.7 | Non-Treatment-Emergent Adverse Events |
|---------------|---------------------------------------------------|
| 16.2.6 | Listing Laboratory Measurements by Subject |
| 16.2.6.1 | Normal Range of Laboratory Values |
| 16.2.6.2 | Hematology (Part I) |
| 16.2.6.3 | Hematology (Part II) |
| 16.2.6.4 | Biochemistry (Part I) |
| 16.2.6.5 | Biochemistry (Part II) |
| 16.2.6.6 | Biochemistry (Part III) |
| 16.2.6.7 | Coagulation |
| 16.2.6.8 | Urinalysis |
| 16.2.6.9 | Urine Microscopy |
| 16.2.6.10 | Pregnancy Test |
| 16.2.6.11 | Additional (Not Planned) Laboratory Safety Tests |
| 16.2.7 | Vital Signs |
| 16.2.7.1 | Vital Signs |
| 16.2.8 | 12-Lead ECG |
| 16.2.8.1 | 12-Lead ECG |
| 16.2.9 | Individual Pharmacokinetic Data |
| 16.2.9.1 | Individual Pharmacokinetic Data |
| 16.2.9.1.1 | Cytisine: Individual Drug Concentration Data |
| 16.2.9.1.2 | Cytisine: Individual Pharmacokinetic Parameters |
| 16.2.9.2 | Documentation of Non-Compartmental Analysis (NCA) |
| 16.2.9.3 | Cytisine: ACH-CYT-08 Phoenix NCA Output |
| 16.2.10 | Concomitant Medication |
| 16.2.10.1 | Concomitant Medication |
| 16.4 INDIVIDU | JAL SUBJECT DATA LISTINGS (US Archival Listings) |

# 10. REFERENCES

[1] ACH-CYT-08 Clinical Study Protocol, Version 5.0, 07MAY2019.

Protocol: ACH-CYT-08 Version: 2.0 Date: 09OCT2019




# 11. APPENDICES

ACH-CYT-08 TFL Date: ddMMMyyyy




# Table A. Study flow-chart

Note: To be captured from the Clinical Study Protocol and Amendments.

# **Table B. Identity of Investigational Products**

Note: To be generated by the MW.

Date: ddMMMyyyy





Date: ddMMMyyyy





ACH-CYT-08 TFL Date: ddMMMyyyy



Date: ddMMMyyyy

Date: ddMMMyyyy





TFL

Date: ddMMMyyyy





Date: ddMMMyyyy





TFL Date: ddMMMyyyy








ACH-CYT-08

Date: ddMMMyyyy






















ACH-CYT-08 TFL Date: ddMMMyyyy









ACH-CYT-08 TFL Date: ddMMMyyyy





ACH-CYT-08 TFL Date: ddMMMyyyy









Date: ddMMMyyyy

















TFL

Date: ddMMMyyyy





Date: ddMMMyyyy



ACH-CYT-08 TFL

Date: ddMMMyyyy


## 14.3. PHARMACOKINETIC DATA





ACH-CYT-08
TFL
Date: ddMMMyyyy



Date: ddMMMyyyy


















































































ACH-CYT-08 TFL

Date: ddMMMyyyy









ACH-CYT-08 TFL Date: ddMMMyyyy















ACH-CYT-08 TFL

Date: ddMMMyyyy




#### 12. ANNEXES

- [1] Data Blind Review Process Minutes 10OCT2019.
- [2] List of Dosed Subjects.



### ACH-CYT-08 Annex 2

### **Annex 2: Data Blind Review Process Minute**








## ACH-CYT-08 Annex 2






# ACH-CYT-08 Annex 2






























Page13 of 13